CLINICAL TRIAL: NCT04872426
Title: Effect of Ischemia on the Insulin-sensitizing Effect of Exercise
Brief Title: Ischemia-reperfusion Exercise Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Professor Jorgen FP Wojtaszewski, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Ischemia
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-04

CONDITIONS: Insulin Sensitivity
Keywords: Exercise; Glucose Uptake; Ischemia; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance; Motor Activity; Ischemia | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low intensity exercise (Experimental): 70% of maximal leg work load capacity
  Interventions: Other: Exercise, insulin infusion
- High intensity exercise (Experimental): 70% and 95% of maximal work load capacity (alternately every 5 min)
  Interventions: Other: Exercise, insulin infusion
- Low intensity exercise + intermittent ischemia-reperfusion (Experimental): 70% of maximal leg work load capacity with intermittent ischemia (25 seconds every 2 min)
  Interventions: Other: Exercise, insulin infusion

INTERVENTIONS:
Other: Exercise, insulin infusion — Acute one-legged exercise, Insulin infusion 3 hours after one-legged exercise

SUMMARY:
The study investigates the relationship between activation of AMP-activated protein kinase (AMPK) in human skeletal muscle and the subsequent improvement in muscle insulin sensitivity for the stimulation of glucose uptake.

This will be investigated in young healthy lean male subjects.

DETAILED DESCRIPTION:
This study aims to demonstrate the association between AMPK activation and increased insulin sensitivity in human skeletal muscle. The investigators intend to examine insulin sensitivity after various levels of AMPK activation in skeletal muscle that includes exercise at different intensities as well as exercise combined with leg blood flow restriction (ischemia). The hypothesis is that exercise combined with ischemia will result in an increased activation of AMPK compared to exercise alone, and therefore it is expected that exercise combined with ischemia will result in the greatest improvement in muscle insulin sensitivity.

Methods:

The main experiment consists of 3 experimental days (A, B and C), separated by a minimum of 14 days and carried out in a randomised order. On all the study days, the participants will arrive in the laboratory after an overnight fast. Catheters will be placed in both femoral veins and in one femoral artery. A muscle biopsy will be obtained from vastus lateralis of one leg (resting leg). Experiment A consists of one-legged muscle work for 1 hour at 70% of the leg maximum aerobic work capacity with the other leg serving as a resting control. In experiment B, the same work are performed, but with periodic at the same constricting the blood supply to the working leg (25 seconds every 2 min). Experiment C consists of one-legged muscle work for 1 hour at 70% and 95% of the leg maximum aerobic work capacity (alternately every 5 min). Immediately after each type of exercise a biopsy will be obtained from the exercising leg and the participants will rest in the fasted state for 3 hours before a third set of muscle biopsies (from both legs) will be obtained. Subsequently, insulin sensitivity will be evaluated in the participants during a 2-hour physiological hyperinsulinemic euglycemic clamp. By the end of the clamp, a final set of biopsies (both legs) will be obtained. Throughout the study day sampling of artery and venous blood/plasma samples allows for the estimation of substrate extraction by the two legs. Further, measures of artery blood flow by Ultrasound Doppler technique allow for the final calculation of substrate uptake/release across the two legs before exercise, during exercise and in recovery from exercise. Importantly, the ability for insulin to stimulate these processes can be evaluated in both a rested and in a prior exercised leg.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (BMI: below or equal to 27)
* physical active on a regular basis
* cardiorespiratory fitness between 40-60 ml/kg/min
* no history or sign of type 2 diabetes, hypertension, insulin resistance or dyslipidemia

Exclusion Criteria:

* smoker
* BMI: above 27
* using any kind of medication

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Muscle glucose uptake during exercise and enhanced insulin sensitivity in recovery from exercise. | Through study completion, an average of 1 year.
  Leg glucose uptake is calculated by the arterial-venous difference i blood glucose concentration multiplied with leg blood flow. Sampling of artery and venous blood samples for blood glucose measurements. Measures of artery blood flow by Ultrasound Doppler technique allows a final calculation of glucose uptake across the legs before exercise, during exercise, in recovery from exercise and with insulin stimulation.

SECONDARY OUTCOMES:
AMPK activity in muscle biopsies | 5 years
  The obtained muscle samples will be subjected to protein kinase activity measurements.
Posttranslational modification of proteins in muscle biopsies | 5 years
  The obtained muscle samples will be subjected to standard western blotting for the evaluation of posttranslational modifications of various proteins involved in glucose metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise, Nutrition and Sports, Faculty of Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided